CLINICAL TRIAL: NCT07401511
Title: A Multicenter, Randomized Controlled Clinical Study Evaluating the Efficacy of Dynamic Spatiotemporal Optical Film (S.T.O.P®KIT) in Retarding Axial Length Growth in Children With Low Hyperopia
Brief Title: Efficacy of S.T.O.P®KIT in Retarding Axial Length Growth in Children With Low Hyperopia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaojuan Wang, Director of the Optometry Department, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20250924101843325
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Children; Hyperopia
Keywords: children; axial length; low hyperopia; spherical equivalent; Dynamic Spatiotemporal Optical Film
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Attaching different phase Dynamic Spatiotemporal Optical Films (S.T.O.P® KIT) when wearing spectacle frames
  Interventions: Device: Attaching different phase Dynamic Spatiotemporal Optical Films (S.T.O.P® KIT) when wearing spectacle frames
- Control group (No Intervention): No active intervention measures

INTERVENTIONS:
Device: Attaching different phase Dynamic Spatiotemporal Optical Films (S.T.O.P® KIT) when wearing spectacle frames — 1. First, two pairs of eyeglasses need to be fitted, with S.T.O.P optical films of different phases attached regularly;
  2. Follow-up visits are conducted every 3 months, and eyeglasses are replaced at 6 months (with changes in S.T.O.P optical film design and phase);
  3. All lenses are plano-spherical and plano-cylindrical lenses (0D sphere, 0D cylinder);
  4. Monitoring of axial length, visual acuity, and corresponding ophthalmic examinations are performed.
  Arms: Experimental Group

SUMMARY:
This is a multicenter, parallel-group, open-label, randomized controlled, superiority interventional clinical study initiated by investigators from Shanghai General Hospital (Study Protocol No.: IT-CRU-FAMB-001, Version V1.1, dated December 29, 2025), with Wang Xiaojuan as the principal investigator and the Department of Ophthalmology as the responsible department, collaborating with The First Affiliated Hospital of Zhengzhou University and Yantai Yuhuangding Hospital as participating centers. Launched on October 1, 2025, and scheduled to complete on April 1, 2027, the study aims to evaluate the efficacy of the Dynamic Spatiotemporal Optical Film (S.T.O.P®KIT) in retarding axial length growth in children with low hyperopia (primary endpoint) and compare the change in spherical equivalent power measured by autorefractometer under cycloplegia between the experimental and control groups (secondary endpoint). A total of 180 eligible children aged 6-10 years with low hyperopia will be randomly divided into the experimental group (90 cases) and the control group (90 cases) at a 1:1 ratio using simple randomization. The experimental group will receive two pairs of customized plano-spherical and plano-cylindrical glasses with S.T.O.P optical films of different phases (replaced at 6 months) and undergo follow-up every 3 months for 12 months, while the control group will only receive regular ophthalmic re-examinations without active intervention (with free dynamic optical films and customized glasses provided upon completion of all follow-ups). The study will adopt Analysis of Covariance (ANCOVA) for statistical analysis, with strict data management and quality control measures in place to ensure data authenticity and reliability, and will comply with the Declaration of Helsinki, Chinese GCP, and relevant ethical requirements to protect the safety, rights, and interests of study participants.

ELIGIBILITY:
Inclusion Criteria:

* Eligible study participants must meet all the following criteria: 1. Age: 6-10 years old;
* +0.75D ≤ Spherical equivalent power ≤ +3.00D;
* Anisometropia ≤ 1.50D;
* Astigmatism ≤ 1.50D;
* No participation in other myopia prevention and control studies or use of other myopia prevention and control methods (including low-concentration atropine eye drops, defocus eyeglasses, orthokeratology lenses, multifocal soft contact lenses, etc.) within 3 months;
* Best-corrected visual acuity (BCVA) in both eyes ≥ 0.8 using a standard logarithmic visual acuity chart;
* Ability to wear frame glasses during near work for at least 6 hours per day;
* Study participants or their legal representatives sign the informed consent form.

Exclusion Criteria:

* Patients with strabismus;
* Patients with abnormal stereopsis;
* Comorbidity with other ophthalmic diseases, including developmental abnormalities affecting visual function and refractive status;
* Previous ocular surgery history;
* Previous receipt of other myopia control treatments (including orthokeratology lenses, multifocal design soft contact lenses or frame glasses, drug therapy [atropine], visual training, etc.);
* Current use of medications that may affect pupil size and ocular surface function;
* Comorbidity with other systemic diseases that may affect visual function or refractive status;
* Family history of hereditary ophthalmic diseases;
* Other conditions deemed unsuitable for participation by investigators.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Difference in the change in axial length | Baseline, 3-month, 6-month, 9-month and 12-month
  Difference in the change in axial length from baseline to 12 months after eyeglass fitting between the experimental group and the control group.

SECONDARY OUTCOMES:
Difference in the change in spherical equivalent power | Baseline, 3-month, 6-month, 9-month and 12-month
  Difference in the change in spherical equivalent power measured by autorefractometer under cycloplegia from baseline to 12 months after eyeglass fitting between the experimental group and the control group.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Zhengzhou University, Zhenzhou, Henan
  - Yuhuangding Hospital of Yantai, Yantai, Shandong
  - Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schmucker C, Lagreze WA. Multifocal Optics for Myopia Control. Klin Monbl Augenheilkd. 2024 Oct;241(10):1129-1133. doi: 10.1055/a-2397-1660. Epub 2024 Oct 9. PMID 39384214
- [Result] Wang M, Ma R, Kuang L, Chen X, Vincent SJ, Tan H, Lai Z, Xu S, Hu Y, Han M, Chen Q, Wang Z, Li L, Yang X. Myopia Control Efficacy of Asymmetric Multipoint Defocus Technique Spectacle Lenses: One-Year Double-Masked Randomized Controlled Trial. Ophthalmology. 2025 Sep;132(9):972-979. doi: 10.1016/j.ophtha.2025.04.022. Epub 2025 Apr 28. PMID 40306584
- [Result] Choi KY, Mok AY, Do CW, Lee PH, Chan HH. The diversified defocus profile of the near-work environment and myopia development. Ophthalmic Physiol Opt. 2020 Jul;40(4):463-471. doi: 10.1111/opo.12698. Epub 2020 Jun 9. PMID 32519412
- [Result] Liu J, Lu Y, Huang D, Yang J, Fan C, Chen C, Li J, Wang Q, Li S, Jiang B, Jiang H, Li X, Yang Z, Lan W. The Efficacy of Defocus Incorporated Multiple Segments Lenses in Slowing Myopia Progression: Results from Diverse Clinical Circumstances. Ophthalmology. 2023 May;130(5):542-550. doi: 10.1016/j.ophtha.2023.01.007. Epub 2023 Jan 13. PMID 36642334
- [Result] Hung GK, Ciuffreda KJ. Incremental retinal-defocus theory of myopia development--schematic analysis and computer simulation. Comput Biol Med. 2007 Jul;37(7):930-46. doi: 10.1016/j.compbiomed.2006.10.004. Epub 2006 Dec 5. PMID 17150204
- [Result] Tang T, Lu Y, Li X, Zhao H, Wang K, Li Y, Zhao M. Comparison of the long-term effects of atropine in combination with Orthokeratology and defocus incorporated multiple segment lenses for myopia control in Chinese children and adolescents. Eye (Lond). 2024 Jun;38(9):1660-1667. doi: 10.1038/s41433-024-02987-5. Epub 2024 Feb 28. PMID 38418604
- [Result] Lembo A, Schiavetti I, Serafino M, Caputo R, Nucci P. Comparison of the performance of myopia control in European children and adolescents with defocus incorporated multiple segments (DIMS) and highly aspherical lenslets (HAL) spectacles. BMJ Paediatr Open. 2024 Dec 31;8(1):e003187. doi: 10.1136/bmjpo-2024-003187. PMID 39741002
- [Result] Lam CSY, Tang WC, Tse DY, Lee RPK, Chun RKM, Hasegawa K, Qi H, Hatanaka T, To CH. Defocus Incorporated Multiple Segments (DIMS) spectacle lenses slow myopia progression: a 2-year randomised clinical trial. Br J Ophthalmol. 2020 Mar;104(3):363-368. doi: 10.1136/bjophthalmol-2018-313739. Epub 2019 May 29. PMID 31142465
- [Result] Fedtke C, Chen Z, Tilia D, Li L, Chen X, Ehrmann K, Lahav-Yacouel K, Falk D, Conrad F, Tan KO, Bakaraju RC. Spatio-Temporal Optical Phase Kit for Myopia Control: Stage 1 Results from a Randomized Controlled Clinical Trial in Chinese Children. Ophthalmology. 2025 Dec;132(12):1344-1356. doi: 10.1016/j.ophtha.2025.08.001. Epub 2025 Aug 7. PMID 40782835

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT07401511/Prot_SAP_000.pdf
  • Informed Consent Form (2025-12-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT07401511/ICF_001.pdf